CLINICAL TRIAL: NCT01456130
Title: A Long-Term, Open-Label Study to Investigate the Long-Term Safety of SYR-322 When Used in Combination With Rapid-Acting Insulin Secretagogues in Subjects With Type 2 Diabetes in Japan
Brief Title: Long-term Study of Alogliptin as an Add-on to Rapid-Acting Insulin Secretagogues in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SYR-322/OCT-901; U1111-1124-8848 (Registry Identifier: WHO); JapicCTI-111643 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-10-13; First posted 2011-10-20 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — alogliptin

ARMS (1):
- Alogliptin (Experimental): Alogliptin 25 mg (or 12.5 mg for participants with moderate renal dysfunction) tablets, orally once daily and a rapid-acting insulin secretagogue as prescribed by the Investigator for up to 52 weeks.
  Interventions: Drug: Alogliptin; Drug: Rapid-acting insulin secretagogue

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322; Nesina®
Drug: Rapid-acting insulin secretagogue — Either of the following commercially available rapid-acting insulin secretagogues as prescribed by the Investigator: (i) Nateglinide: Dose: 30 mg tablet or 90 mg tablet (ii) Mitiglinide calcium hydrate: Dose: 5 mg tablet or 10 mg tablet

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of alogliptin as an add-on to a rapid-acting insulin secretagogue (medicine that stimulates insulin release) in type 2 diabetic patients with inadequate blood glucose control despite treatment with a rapid-acting insulin secretagogue as well as diet and exercise therapies.

DETAILED DESCRIPTION:
One alogliptin 25 mg tablet was orally administered once daily before breakfast for up to 52 weeks.

The dose of alogliptin was adjusted according to the severity of the participant's renal dysfunction based on serum creatinine (SCr) levels. Participants with moderate renal dysfunction (SCr, >1.4 - ≤2.4 mg/dL for men and >1.2 - ≤ 2.0 mg/dL for women) received alogliptin 12.5 mg tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus.
2. Had an HbA1c of ≥ 6.5% and < 10.0% at the start of the observation period (Week -2).
3. Had been receiving specific diet and exercise (if applicable) therapies since at least 10 weeks prior to the start of the observation period (Week -2).
4. Had been receiving basic diabetes treatment with a rapid-acting insulin secretagogue (nateglinide or mitiglinide calcium hydrate) alone using a stable dosage regimen since at least 10 weeks prior to the start of the observation period (Week -2).
5. Was suitable for combination therapy of either of the above rapid-acting insulin secretagogues (nateglinide or mitiglinide calcium hydrate) and another antidiabetic drug at the start of the observation period (Week -2) in the investigator's or subinvestigator's opinion.
6. Participants complicated by hypertension had stable blood pressure control and needed neither dose adjustment of the ongoing antihypertensive (including discontinuation and interruption) nor additional use of another antihypertensive throughout the duration of the study in the investigator's or subinvestigator's opinion.
7. Male or female and aged 20 years or older at the time of signing of informed consent.
8. If female, and of child-bearing potential and sexually active with a nonsterilized male partner agreed to use adequate contraception routinely from signing of informed consent throughout the duration of the study.
9. Visited the study site on an outpatient basis during the observation period.
10. Was capable of understanding and complying with protocol requirements in the investigator's or subinvestigator's opinion.
11. Signed and dated the informed consent documents prior to the start of any study procedures.

Exclusion Criteria:

1. Severe renal dysfunction or end-stage renal disease [e.g., a serum creatinine (SCr) level of >2.4 mg/dL (men) or >2.0 mg/dL (women) at the start of the observation period (Week -2)].
2. Obvious clinical manifestations of hepatic impairment [e.g., an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) value of ≥ 2.5 times the upper limit of normal at the start of the observation period (Week -2)].
3. Any serious cardiac disease, serious cerebrovascular disorder, or serious pancreatic or hematological disease (e.g., requiring hospitalization for treatment).
4. Systolic blood pressure of ≥ 180 mmHg or diastolic blood pressure of ≥ 110 mmHg during the observation period.
5. A condition requiring insulin for blood glucose control (e.g., a patient with severe ketosis, diabetic coma or precoma, type 1 diabetes mellitus, severe infection, a pre- or post-operative condition, or serious trauma).
6. Malignant tumor.
7. History of hypersensitivity or allergies to dipeptidyl-peptidase-4 (DPP-4) inhibitors.
8. A habitual drinker whose daily alcohol consumption was >100 mL on average.
9. A history of drug abuse (defined as any illicit drug use) or alcohol abuse.
10. Required to take excluded medications during the duration of the study.
11. Previously received SYR-322 or Nesina® Tablets in a clinical study or as a therapeutic drug.
12. Received any investigational product (including investigational products for postmarketing clinical studies) within 12 weeks prior to the start of the observation period.
13. Had participated in another clinical study at signing of informed consent.
14. If female, was pregnant or lactating, or intended to become pregnant between signing of informed consent and 1 month after the end of the study; or intended to donate ova during such time period.
15. A study site employee, an immediate family member of a study site employee or in a dependent relationship with a study site employee who was involved in the conduct of this study (e.g., spouse, parent, child, sibling), or might consent under duress.
16. Changed the dosing regimen of the ongoing rapid-acting insulin secretagogue during the observation period.
17. History of hypersensitivity or allergies to rapid-acting insulin secretagogues.
18. Any condition for which Nesina® Tablets, nateglinide, or mitiglinide calcium hydrate was contraindicated as defined in their package inserts.
19. Otherwise ineligible for participation in the study in the investigator's or subinvestigator's opinion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (14):
- Japan (14):
  - Nagoya, Aichi-ken
  - Fukuoka, Fukuoka
  - Kurume-shi, Fukuoka
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Kagoshima, Kagoshima-ken
  - Kumamoto, Kumamoto
  - Osaki-shi, Miyagi
  - Minou-shi, Osaka
  - Osaka, Osaka
  - Kamio-shi, Saitama
  - Koshigaya-shi, Saitama
  - Adachi-ku, Tokyo
  - Chuo-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in Japan from 10 November 2011 to 16 March 2013.
Pre-assignment Details: Patients with type 2 diabetes with inadequate blood glucose control despite treatment with a rapid-acting insulin secretagogue as well as diet and exercise therapies were enrolled in a single treatment group.
Period: Overall Study
Arm/Group | Alogliptin
Started | 67
Completed | 57
Not Completed | 10
Not completed — Adverse Event | 4
Not completed — Voluntary Withdrawal | 1
Not completed — Lack of Efficacy | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alogliptin
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.52)
Age, Customized [Number; unit: participants]
  < 65 years | 37
  ≥ 65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 41
Weight [Mean (Standard Deviation); unit: kg] | 66.64 (14.409)
Height [Mean (Standard Deviation); unit: cm] | 161.7 (10.22)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.38 (4.347)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 7.44 (5.872)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent glycosylated hemoglobin] | 7.63 (0.957)
Baseline hemoglobin A1c (HbA1c) categories [Number; unit: participants]
  < 6.5 % | 3
  ≥ 6.5 and < 7.0% | 17
  ≥ 7.0 and < 8.0% | 25
  ≥ 8.0% | 22
Fasting blood glucose [Mean (Standard Deviation); unit: mg/dL] | 182.1 (45.07)
Fasting blood glucose categories [Number; unit: participants]
  < 130 mg/dL | 6
  ≥ 130 to < 160 mg/dL | 17
  ≥ 160 mg/dL | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An TEAE is any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have a causal relationship with this treatment. A serious TEAE is defined as any untoward medical occurrence that resulted in death, was life threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability or incapacity, led to a congenital anomaly/birth defect or was an important medical event that may have required intervention to prevent any of items above.
Time Frame: 52 Weeks
Population: Safety analysis set - All participants who received at least one dose of the investigational product (alogliptin) and a rapid-acting insulin secretagogue.
Measure: Number; unit: participants
Arm/Group | Alogliptin
Number analyzed (Participants) | 67
participants
  Any adverse event | 57
  Adverse event leading to discontinuation | 5
  Serious adverse event (SAE) | 6
  SAE leading to discontinuation | 0
  Death | 0

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin collected at Week 52 or at the final visit relative to Baseline.
Time Frame: Baseline and Week 52
Population: Full analysis set: All randomized participants who received at least one dose of double-blind study medication.
Measure: Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin
Number analyzed (Participants) | 67
percentage of glycosylated hemoglobin | -0.46 [-0.690 to 0.221]

3. Secondary Outcome: Percentage of Participants With a Clinical Response
Description: Clinical response is defined as an HbA1c level less than 5.8% or less than 6.5% at Week 52 or at the final visit.
Time Frame: Week 52
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alogliptin
Number analyzed (Participants) | 67
percentage of participants
  HbA1c of < 5.8% | 4.5 [0.933 to 12.533]
  HbA1c of < 6.5% | 28.4 [18.015 to 40.691]

4. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: The change in the value of fasting glucose collected at Week 52 or the final visit relative to Baseline.
Time Frame: Baseline and Week 52
Population: Full analysis set.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Alogliptin
Number analyzed (Participants) | 67
mg/dL | -10.5 [-18.75 to -2.30]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin
Serious Adverse Events (participants affected / at risk) | 6/67
Other Adverse Events (participants affected / at risk) | 57/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin (N=67)
Bronchiolitis (Infections and infestations) | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myocardial infarction (Cardiac disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin (N=67)
Nasopharyngitis (Infections and infestations) | 24
Bronchitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Periodontitis (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 2
Seasonal allergy (Immune system disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 2
Headache (Nervous system disorders) | 3
Asthenopia (Eye disorders) | 3
Cataract (Eye disorders) | 2
Conjunctivitis allergic (Eye disorders) | 2
Diabetic retinopathy (Eye disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Dental caries (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Diabetic nephropathy (Renal and urinary disorders) | 4
Chest pain (General disorders) | 2
Malaise (General disorders) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.